CLINICAL TRIAL: NCT01955629
Title: A Single-Arm, Open Label Study of Aflibercept as Maintenance Therapy Following Induction With Aflibercept in Combination With XELOX, as First-Line Treatment for Metastatic Colorectal Cancer Patient
Brief Title: Study of Aflibercept as Maintenance Therapy Following Induction With Aflibercept in Combination With XELOX, as First-Line Treatment for Metastatic Colorectal Cancer Patient
Acronym: AMOR
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study enrollment was prematurely halted due to safety reasons.
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFLIBC06561; 2013-000858-22; U1111-1143-3015 (Other: UTN)
Record Dates: First submitted 2013-09-13; First posted 2013-10-07 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — aflibercept; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept + XELOX (Oxaliplatin and Capecitabine) (Experimental): Aflibercept 6 mg/kg every 3 weeks (q3w) in combination with Oxaliplatin 100 mg/m^2 q3w and Capecitabine 850 mg/m^2 twice daily orally (from Day 1 to Day 14 of each cycle), up to 6 cycles as induction therapy, followed by aflibercept 6 mg/kg q3w as maintenance therapy up to disease progression or unacceptable toxicity or participant's refusal of further treatment.
  Interventions: Drug: Aflibercept AVE0005; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Aflibercept AVE0005 — Pharmaceutical form: Concentrate for solution for infusion; Route of administration: Intravenous
  Other Names: Zaltrap
Drug: Oxaliplatin — Pharmaceutical form: Concentrate for solution for infusion; Route of administration: Intravenous
  Other Names: Eloxatin; SR96669
Drug: Capecitabine — Pharmaceutical form: Tablets; Route of administration: Oral

SUMMARY:
Primary Objectives:

Study Part 1: To determine the recommended dose for the aflibercept, oxaliplatin and capecitabine (XELOX) combination to be used in the Part 2 of the study.

Study Part 2: To assess the percentage of participants without progression of the disease at 6 months after the start of maintenance therapy with aflibercept single-agent, following the first-line induction therapy with XELOX and aflibercept combination in participants with previously untreated metastatic colorectal cancer.

Secondary Objective:

Study Part 2: Include the evaluation of progression free survival, overall survival, response to treatment, the overall safety (during induction and maintenance therapy) and the assessment of aflibercept pharmacodynamics and biomarkers parameters.

DETAILED DESCRIPTION:
The duration of the study for each participant includes a period for screening of up to 3 weeks, study drug administrations every 3 weeks up to disease progression, unacceptable toxicity or participant's refusal of further study treatment, followed by a minimum of 30-day follow-up after the last study treatment administration.

After study treatment discontinuation each participant will be followed-up until death, participant's refusal or end of study (whichever comes first).

This trial is being conducted in Europe, where the INN designation for the study molecule is "aflibercept" and this term is therefore used throughout the synopsis. In the US, the US proper name is "ziv-aflibercept".

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically-proven adenocarcinoma of the colon or rectum.
* Metastatic disease not amenable to potentially curative treatment (i.e. unresectable).
* Measurable lesion as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* No prior systemic anti-cancer treatment for metastatic disease.
* No prior adjuvant treatment after resection of distant metastases.
* No prior treatment with angiogenesis inhibitors.

Exclusion criteria:

* Age <18 years.
* Eastern Cooperative Oncology Group Performance status >/= 2.
* Less than 4 weeks from prior radiotherapy or prior surgery (or until the surgical wound is fully healed).
* Treatment with any other investigational product within the prior 28 days.
* Other prior neoplasm.
* History of brain metastases, active seizure disorder, uncontrolled spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease.
* Any of the following within the prior 6 months: myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, severe congestive heart failure, stroke or transient ischemic attack.
* Any of the following within the prior 3 months: moderate/severe gastrointestinal bleeding/hemorrhage, treatment resistant peptic ulcer disease, erosive oesophagitis or gastritis, infectious or inflammatory bowel disease, diverticulitis, pulmonary embolism or other uncontrolled thromboembolic event.
* Deep vein thrombosis within the prior 4 weeks.
* Any severe acute or chronic medical condition, which could impair the ability of the participant to participate in the study.
* Inadequate bone marrow, liver and renal function: neutrophils < 1.5x10^9/L, platelets < 100x10^9/L, hemoglobin < 9.0 g/dL, total bilirubin >1.5 x upper normal limit (ULN), transaminases >3 x ULN (unless liver metastasis are present), alkaline phosphatase >3 x ULN (unless liver metastasis are present), serum creatinine > 1.5 x ULN.
* Participants on anticoagulant therapy with warfarin.
* Symptomatic peripheral sensory neuropathy.
* Inability to take oral medications.
* Prior history of chronic enteropathy, inflammatory enteropathy, chronic diarrhea, malabsorption syndrome, unresolved bowel obstruction/sub-obstruction, surgery more extensive than hemicolectomy, extensive small intestine resection with chronic diarrhea.
* Known dihydropyrimidine dehydrogenase deficiency.
* known history of hypersensitivity to aflibercept.
* Any contraindication to administer oxaliplatin or capecitabine as per package insert of each drug.
* Urine protein-creatinine ratio (UPCR) >1 on morning spot urinalysis or proteinuria > 500 mg/24-h.
* Uncontrolled hypertension within the prior 3 months.
* Evidence of clinically significant bleeding predisposition or underlying coagulopathy, non-healing wound.
* Pregnant or breast-feeding women.
* Participants with reproductive potential who do not agree to use an accepted effective method of contraception.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Italy (2):
  - Investigational Site Number 380-001, Genova
  - Investigational Site Number 380-002, Milan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 sites in Italy. A total of 6 participants were screened between 17 Dec 2013 and 24 Feb 2014, out of which 4 participants were enrolled and treated.
Pre-assignment Details: Participants enrolled in Part-1 of study to assess recommended phase 2 dose (RP2D) of combination of aflibercept with oxaliplatin and capecitabine. 3 participants discontinued due to adverse events (AE) and 1 participant due to disease progression (DP) at dose level 1 of treatment. Part-2 of study (efficacy and safety evaluation) was not performed.
Groups:
- Aflibercept + XELOX (Oxaliplatin and Capecitabine): Aflibercept 6 mg/kg intravenous (IV) infusion every 3 weeks (q3w) in combination with Oxaliplatin 100 mg/m^2 IV infusion q3w and Capecitabine 850 mg/m^2 twice daily orally (from Day 1 to Day 14 of each cycle), up to 6 cycles as induction therapy, followed by aflibercept 6 mg/kg IV infusion q3w as maintenance therapy up to DP or unacceptable toxicity or participant's refusal of further treatment.
Period: Overall Study
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Started | 4
Completed | 4 (1 participant with DP and 3 with unacceptable toxicity were considered completed as per protocol.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Aflibercept + XELOX (Oxaliplatin and Capecitabine): Aflibercept 6 mg/kg IV infusion q3w in combination with Oxaliplatin 100 mg/m^2 IV infusion q3w and Capecitabine 850 mg/m^2 twice daily orally (from Day 1 to Day 14 of each cycle), up to 6 cycles as induction therapy, followed by aflibercept 6 mg/kg IV infusion q3w as maintenance therapy up to DP or unacceptable toxicity or participant's refusal of further treatment.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were assessed using the national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) version 4.03. DLTs were defined as any of following AEs: grade 4 neutropenia lasting >7 consecutive days; febrile neutropenia or neutropenic infection; grade 4 thrombocytopenia; grade 3 thrombocytopenia associated with bleeding requiring transfusion; grade 4 non-hematological treatment related event; grade 3 nausea/vomiting or diarrhea lasting >/= 4 days despite corrective measures; grade 3 other non-hematological toxicities: anorexia, fatigue, hypertension only if G4 or not medically controlled and G3 peripheral sensory neuropathy that did not improve to G<2 at time of retreatment; urinary protein excretion of >3.5 gram per 24 hours that did not recover to <2.0 gram per 24 hours within 2 weeks; symptomatic arterial thromboembolic events including cerebrovascular accidents, myocardial infarction, transient ischemic attacks, new onset or worsening of pre-existing angina.
Time Frame: Cycle 1 (Up to 3 weeks)
Population: Evaluable DLT population defined as the subset of the whole part 1 participants that were exposed to at least 1 dose (even incomplete) of the study treatment and had a DLT assessment at Cycle 1.
Measure: Number; unit: Participants
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 4
Participants | 1

2. Primary Outcome: Part 2: Number of Participants With Progression Free Survival (PFS) at 6 Months After the Start of Maintenance Therapy
Description: It describes the number of participants alive without progression at 6 months after the start of Aflibercept maintenance therapy.
Time Frame: 6 months after the start of maintenance therapy.
Population: Due to premature recruitment discontinuation, none of the planned efficacy analyses was performed.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 0

3. Secondary Outcome: Part 1: Number of Participants With Tumor Responses (Complete Response [CR], Partial Response [PR], Stable Disease [SD] or Progressive Disease [PD])
Description: Tumor assessment was performed by abdomino-pelvic computed tomography scan or magnetic resonance imaging (MRI) and chest X-ray or chest CT-scan to assess the disease status at baseline and then every 9 weeks during study treatment up to DP. Target lesions were evaluated using response evaluation criteria in solid tumors (RECIST) version 1.1, wherein CR = disappearance of all target lesions; PR = 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD; PD =20% increase in the sum of the LD of target lesions taking as reference the smallest sum in the study and SD = small changes that did not meet above criteria.
Time Frame: Baseline and every 9 weeks up to DP (up to 15 months).
Population: Evaluable Population (EP) for tumor response was defined as a subset of ITT population (all participants who gave their informed consent and successfully registered into study) with measurable disease at study entry, who received at least 1 cycle of study treatment, with at least 1 post baseline tumor evaluation, except for early DP or death.
Measure: Number; unit: Participants
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 4
Participants
  CR | 0
  PR | 1
  PD | 0
  SD | 3

4. Secondary Outcome: Part 2: Progression Free Survival (PFS)
Description: PFS was defined as the time interval from the date of registration into the study to the date of first observation of DP or death (due to any cause), whichever was first.
Time Frame: From the date of enrollment up to the date of DP or death, whichever occurred first (up to 15 months).
Population: Due to premature recruitment discontinuation, none of the planned efficacy analyses was performed.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 0

5. Secondary Outcome: Part 2: Overall Survival (OS)
Description: OS was defined as the time interval from the date of registration into the study to the date of death due to any cause. In the absence of confirmation of death, survival time was to be censored at the earliest between the last date the participant was known to be alive and the end of study date.
Time Frame: From the date of enrollment up to the date of death (up to 15 months).
Population: Due to premature recruitment discontinuation, none of the planned efficacy analyses was performed.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 0

6. Secondary Outcome: Part 2: Overall Rate of Resectability of Metastatic Lesions
Description: Overall metastases resection rate was defined as the percentage of participants reaching an R0 metastases resection, defined as the complete absence of invasive carcinoma on histological examination at the time of definitive surgery.
Time Frame: 12 months after the last participant enrolled.
Population: Due to premature recruitment discontinuation, none of the planned efficacy analyses was performed.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 0

7. Secondary Outcome: Part 2: Number of Participants With CR or PR
Description: Tumor assessment was performed by abdomino-pelvic computed tomography scan or MRI and chest X-ray or chest CT-scan to assess the disease status at baseline and then every 9 weeks during study treatment up to DP. Target lesions were evaluated using RECIST version 1.1, wherein CR = disappearance of all target lesions; PR = 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
Time Frame: Baseline and every 9 weeks up to end of study completion (15 months).
Population: Due to premature recruitment discontinuation, none of the planned efficacy analyses was performed.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 0

8. Secondary Outcome: Part 2: Pharmacodynamic Parameters: Modulation of Circulating Analytes
Description: Blood and tumor samples were to be collected to evaluate the pharmacodynamic parameters including the assessment of the modulation of circulating analytes such as cytokines and angiogenic factors.
Time Frame: Baseline (within 21 days before registration); Day 1/pre-dose of Cycle 1, 2 and 3 of induction phase and maintenance phase; 30 ± 3 days after the last aflibercept administration.
Population: Due to premature recruitment discontinuation, no samples had been collected and none of the planned efficacy/pharmacodynamic analyses was performed.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 0

9. Secondary Outcome: Part 2: Aflibercept Biomarkers Evaluation
Description: Blood and tumor samples were to be collected to evaluate proteomic biomarkers such as factors and receptors related to angiogenesis process, inflammation, and tumor progression.
Time Frame: as for outcome 8
Population: Due to premature recruitment discontinuation, no samples had been collected and none of the planned biomarker analyses was performed.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from signature of the informed consent form up to 30 days after the last administration of treatment regardless of seriousness or relationship to study treatment.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (from the first study treatment administration to 30 days after the last study treatment administration).
Groups:
- Aflibercept + XELOX (Oxaliplatin and Capecitabine): Aflibercept 6 mg/kg intravenous(IV) infusion every 3 weeks (q3w) in combination with Oxaliplatin 100 mg/m^2 IV infusion q3w and Capecitabine 850 mg/m^2 twice daily orally (from Day 1 to Day 14 of each cycle), up to 6 cycles as induction therapy, followed by aflibercept 6 mg/kg IV infusion q3w as maintenance therapy up to DP or unacceptable toxicity or participant's refusal of further treatment.
Arm/Group | Aflibercept + XELOX (Oxaliplatin and Capecitabine)
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + XELOX (Oxaliplatin and Capecitabine) (N=4)
Acute coronary syndrome (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Hypertension (Vascular disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aflibercept + XELOX (Oxaliplatin and Capecitabine) (N=4)
Bradycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Localised oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Device related infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study enrollment was prematurely halted due to safety reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.